CLINICAL TRIAL: NCT04854005
Title: Selective Use of ALND in N1 HR+/HER2- Breast Cancer Patients With 1 or 2 Positive Sentinel Lymph Nodes Undergoing Upfront Breast Surgery and Adjuvant Radiation: A Prospective Study
Brief Title: Use of Sentinel Lymph Node Biopsy in Patients With Early-Stage, Palpable Node-Positive HR+/HER2- Breast Cancer Having Upfront Surgery and Adjuvant Radiation
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-183
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Sentinel Lymph Node Biopsy; Palpable Node-Positive HR+/HER2; 21-183
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer: Patients with cTx/cT1-2cN1 HR+/HER2- tumors who are scheduled to undergo upfront surgery will undergo AUS at the enrolling institution to characterize suspicious-appearing lymph nodes, as is part of routine practice.
  Interventions: Procedure: Breast surgery

INTERVENTIONS:
Procedure: Breast surgery — Patients will undergo SLNB with single or dual-tracer lymphatic with technetium-99m sulfur colloid either lymphazurin or methylene blue dye, per institution standard, in accordance with routine clinical practice.

SUMMARY:
The purpose of this study is to find out how often the researchers can avoid an ALND in patients with early-stage, node-positive HR+/HER2- breast cancer who are having upfront surgery. The study researchers think that, if AUS before surgery can help identify people who may have up to 3 affected lymph nodes, it will be possible to perform the less radical standard SLNB during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with biopsy-proven invasive breast cancer
* Patients with cTx, cT1, or cT2 tumors with palpable ipsilateral mobile adenopathy of level I/II axillary nodes with biopsy-proven (either by pre-operative biopsy or intraoperative frozen section) nodal metastasis (cN1) who are undergoing upfront surgery
* Patients with tumors of the HR+/HER2- subtype, defined as:

  1. HR+: Positive for estrogen receptor and/or progesterone receptor staining, indicated by ≥1% immunoreactive tumor nuclei
  2. HER2-: Immunohistochemistry assay demonstrating no or faint staining in ≤10% of tumor cells (IHC 0 or 1+) or negative by dual probe in situ hybridization assay

Exclusion Criteria:

* Patients with prior ipsilateral breast cancer
* Patients who are pregnant
* Patients with stage IV disease at presentation
* Patients with advanced regional disease (cN2/cN3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the Principal Investigator (PI), or the research team at MSKCC/participating institutions.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
evaluate rates of axillary lymph node dissection | 2 years
  Completion ALND will be required if metastases are present in ≥3 SLNs on pathologic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Mamtani, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Hartford Healthcare Cancer Alliance (Data collection only), Hartford, Connecticut
  - University of Michigan (Data Collection Only), Ann Arbor, Michigan
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York
  - Lehigh Valley Health Network (Dara Collection Only), Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm